CLINICAL TRIAL: NCT01235273
Title: Phase 2 Study of Growth Hormone Administration in Patients With Chronic Heart Failure and Low IGF-1 Levels
Brief Title: Treatment of the lOw IGF-1 Syndrome aSsociated With Chronic Heart fAilure: A Randomized, Placebo-Controlled, Double-Blind Study.
Acronym: TOSCA2
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Cittadini, Associate Professor of Internal Medicine, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOSCAproject
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GH replacement therapy (Experimental)
  Interventions: Drug: Growth Hormone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Growth Hormone — growth hormone administration
  Arms: GH replacement therapy
Other: Placebo — standard placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to determine whether treatment of the low IGF-1 syndrome in patients with CHF is able to modify some functional parameters, recognized as valid surrogate end-points of CHF progression.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex affected by CHF NYHA class II-III, secondary to ischemic or idiopathic dilated cardiomyopathy
* age range 30-80 years
* stable medications for at least two months prior to randomization, including ACE inhibitors or AT1 antagonists and beta-blockers (unless untolerated).
* LV ejection fraction 40% or less
* Peak VO2 consumption during a CPET ≤ 16 ml/kg/min.
* LV end-diastolic dimension 55 mm or more
* low IGF-1 levels and a satisfactory response to an IGF-1 generation test
* informed consent

Exclusion Criteria:

* haemodynamic clinically significant primary valvular disease or significant congenital heart disease
* acute pericarditis/myocarditis
* inability to perform a bicycle exercise test
* Poorly controlled diabetes mellitus (HbA1c >8.5)
* active proliferative or severe non-proliferative diabetic retinopathy
* active and/or history of malignancy
* evidence of progression or recurrence of an underlying intracranial tumor
* unstable angina or recent myocardial infarction (less than 5 months)
* severe liver disease
* serum creatinine levels >2.5 mg/dl
* Inability to cooperate or administer the study drug
* Patients participating in any other clinical study, within 30 days prior to screening visit and/or during this particular study period

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
increase of peak VO2 consumption by at least 2.5 ml/kg/min during maximal physical exercise test. | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Cittadini, Napoli, Italy